CLINICAL TRIAL: NCT00815243
Title: Study of Clinical Workflow Changes, Anatomical and Functional Outcomes Due to Telemedicine Consultations in Trauma and Orthopedic
Brief Title: Telemedicine Consultation in Trauma and Orthopedic
Acronym: TeleTO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Donetsk National Medical University (Other)
Responsible Party: Anton Vladzymyrskyy, M.D., Head of Dep. of Informaics and Telemedicine, Donetsk R&D Institute of Traumatology and Orthopedics
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-2007-2011
Record Dates: First submitted 2008-12-26; First posted 2008-12-29 (Estimated); Last update posted 2008-12-29 (Estimated); Status verified 2008-12

CONDITIONS: Trauma; Congenital Bone and Joint Abnormalities; Joint Diseases; Orthopedic Surgery Complications
Keywords: fracture; coxarthrosis; complication; congenital abnormalities; bone; joint; telemedicine; transportation; decision making; outcomes
MeSH Terms: conditions — Wounds and Injuries; Joint Diseases; Fractures, Bone; Osteoarthritis, Hip; Congenital Abnormalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Telemed (Experimental): Group of trauma&orthopedic patients - for determination of clinical strategy and treatment plan telemedicine will be used
  Interventions: Procedure: Telemedicine consultation; Procedure: Treatment plan
- InternalControl (Active Comparator): Group of trauma&orthopedic patients from 3rd level trauma center - for determination of clinical strategy and treatment plan usual clinical approaches will be used
  Interventions: Procedure: Treatment plan
- ExternalControl (Active Comparator): Group of trauma&orthopedic patients from 1-2rd level trauma centers (in rural and small municipal hospitals) - for determination of clinical strategy and treatment plan personal arriving of the expert by the car (so-called Urgent Expert Care) will be used
  Interventions: Procedure: Treatment plan

INTERVENTIONS:
Procedure: Telemedicine consultation — Standard synchronous or asynchronous telemedicine consultations according recommendations and best practice models of ISfTeH
  Other Names: Telemedicine work station according national recommendations; Best practice models for teletrauma recognised by ISFTEH
  Arms: Telemed
Procedure: Treatment plan — Treatment plan include diagnostic tests (physical examination, laboratory tests, xray, CT, MRI), medications and surgical treatment (debridements, osteosynthesis, arthroplasty, ORIF etc)
  Other Names: Ilizarov frame; AO-Plate osteosynthesis; Intermedullar nailing; Total cemented/uncemented hip arthroplasty

SUMMARY:
The purpose of this study is to determine whether telemedicine consultations (lead by standard scheme)allows to increase quality of anatomical and functional outcomes and improve clinical work-flow at patients with acute bone and joint trauma, hip pathology and congenital orthopedics abnormalities.

DETAILED DESCRIPTION:
Levels of bad outcomes, untimely death and disability due to acute trauma, specific orthopedic pathology (congenital, coxarthrosis) and non-efficient organisation of clinical work-flow are still very high (especially in rural areas). Standard telemedicine work stations (with special protocols and manuals for original approach to telemedicine activity organisation and management) will be placed into small municipal and rural hospitals. Telemedicine links will be established between 3rd level Trauma&Ortho center and remote sites. Synchronous and asynchronous teleconsultations will be perform for help in evidence-based timely clinical decisions, continual support of clinical wor-flow and treatment process.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of injury of locomotorium (isolated or polytrauma)
* Clinical diagnosis of bone and joint congenital abnormalities or intranatal injury
* Clinical diagnosis of knee, hip arthrosis
* Clinical diagnosis of complication of surgery (unstable, fracture of construction etc)
* Diagnosis is already present
* Primary decision of clinical strategy have to be done (transportation, level of care, method of treatment, surgery peculiarities)
* Indications for teleconsultations determined by physician

Exclusion Criteria:

* Diagnosis is not present
* Patient's self-request for teleconsultations
* No reliable feed-back with attending physician

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2007-09; Primary Completion 2008-04 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
Scales for outcomes in trauma and orthopedic (Harris Hip Score, national protocol for trauma outcomes). Sets of criteria: ARR, RRR, ABІ, RBI, RR, odds ratio and NNT | one year

SECONDARY OUTCOMES:
"Relevance of Telemedicine Consultation" Questionnaire | one year

CONTACTS AND LOCATIONS:
Overall Officials: Anton V Vladzymyrskyy, M.D., Principal Investigator — R&D Institute of Traumatology and Orthopedics; Volodymyr G Klymovytskyy, Professor, Study Director — R&D Institute of Traumatology and Orthopedics
Locations (5):
- Ukraine (5):
  - Volnovakha Central Area Hospital, Volnovakha, Donetsk Oblast
  - Gorlovka Municipal Hospital N2, Gorlovka, Donetskya Oblast
  - Central Clinical Municipal Hospital N6, Donetsk
  - Donetsk R&D Institute of Traumatology and Orthopedics, Donetsk
  - Clinics of Maxillo-Fascial Surgery of DNMU, Donetsk

REFERENCES:
- [Background] Vladzymyrskyy AV. Four years' experience of teleconsultations in daily clinical practice. J Telemed Telecare. 2005;11(6):294-7. doi: 10.1258/1357633054893337. PMID 16168165
- [Background] Vladzymyrskyy AV. Our experience with telemedicine in traumatology and orthopedics. Ulus Travma Acil Cerrahi Derg. 2004 Jul;10(3):189-91. PMID 15286891
- See also: Best Practice Models in Telemedicine for Trauma (recognized by ISFTEH) — http://www.isft.net/cms/index.php?gpm_best_practice_models
- See also: Med-e-Tel Digital Library: 2005-2007 presentations and papers about telemedicine activity of investigators — http://www.medetel.lu/index.php?rub=library_country&page=ukraine